CLINICAL TRIAL: NCT04293315
Title: Evaluation of the Effectiveness of a Collaborative Strategy to Increase the Screening of Colorectal Cancer in the Public Healthcare Sector in Argentina
Brief Title: Screening of Colorectal Cancer in the Public Healthcare Sector in Argentina
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Institute for Clinical Effectiveness and Health Policy (Other)
Collaborators: Inter-American Development Bank (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: BID CCR
Record Dates: First submitted 2020-01-31; First posted 2020-03-03 (Actual); Last update posted 2020-03-03 (Actual); Status verified 2019-04

CONDITIONS: Colorectal Neoplasms
Keywords: screening; Fecal Occult Blood Test (FOBT); prevention; quality improvement cycles; health promotion
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: Pragmatic Cluster Randomized Controlled Trial. Implementation Hybrid Type 2 Study. It will be used:
  Process Model: CFIR Theory of Change: COM-B Evaluation Framework: RE-AIM
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): This is the usual care arm. Healthcare workers will provide people with the Fecal Occult Blood Test (FOBT) and information about risk to develop CRC and the importance of early detection.
- Intervention (Experimental): The same as the Control Arm plus the primary care team of the PCCs will be trained and participate in 8 improvement cycles.
  Interventions: Behavioral: Improvement Cycles

INTERVENTIONS:
Behavioral: Improvement Cycles — This is a multi-component intervention following the Institute for Healthcare Improvement (IHI)'s Collaborative Model for Achieving Breakthrough Improvement by implementing "plan-do-study-act" (PDSA) improvement cycles. The investigators will conduct 8 participative learning sessions for the primary care team. These sessions will be aimed at identifying opportunities for improvement oriented to the design and application of innovative approaches based on best practices.
  Other Names: quality improvement cycle
  Arms: Intervention

SUMMARY:
Introduction: Early detection of certain types of cancer significantly increases the likelihood of successful treatment and reduces mortality from these causes. However, the use of screening and the early detection of selected tumors such as colorectal cancer (CRC) are lower than those expected in our country. The objective of this project is to evaluate the effectiveness of a multicomponent strategy that improves the screening and early detection of CRC in the population at risk of Primary Health Care Clinics (PCCs) of the public health system.

Population: people leaving in the catchment area of 10 selected primary care clinics from the public health system in the province of Mendoza, Argentina.

Design and methods: a Randomized clinical study by clusters. 10 PCCs will be included: 5 will be randomly assigned to receive an intervention to increase the CRC screening rates (improvement cycles) and 5 to the control arm (usual care). 150 participants will be included in each PCCs, in total, 1500 participants.

Intervention: An innovative vision is proposed, which combines a participatory and dynamic methodology based on improvement cycles. This approach includes the implementation of participatory learning sessions for health providers, involving the effectors of the design of the intervention. In the intervention branch at least 3 workshops (sessions) will be held with the members of the care system, in order to identify opportunities for improvement oriented to the design and application of an innovative intervention based on best practices. Each one of the sessions will constitute an analysis of the improvement cycle, following the following steps: 1) Selection of participants of the initial workshop; 2) Development of work model based on bibliographic review and initial qualitative phase; 3) Initial workshop with effectors for training in continuous improvement, objectives, interventions and data collection; 4) Learning workshops to discuss results, applicability of interventions and modifications to the work plan; 5) Closing session to evaluate preliminary results and discuss continuity of interventions beyond the project.

Outcomes: 1) Percentage of the population at risk that completes the screening; 2) Percentage of the population classified as at habitual risk or increased by risk factors.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have public health coverage
* Age between 50 and 75 years old
* Residence in the catchment area of the PCCs
* With an indication to perform screening for CRC with FOBT
* People who consent to participate

Exclusion Criteria:

* People who are bedridden.
* People who plan to move in the next 3 months.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1520 (Actual)
Dates: Start 2018-06-09 (Actual); Primary Completion 2020-03-15 (Estimated); Study Completion 2020-03-15 (Estimated)

PRIMARY OUTCOMES:
Effective Screening | 3 months
  Proportion of participants who with known result of the FOBT within 90 days from recruitment. The investigators will review National Information System Registry to count the number of participants in each arm with a known result for their FOBT. The investigators will calculate the proportion of participants with known result (Effective Screening) in each arm of the study.

SECONDARY OUTCOMES:
Proportion of participants with inadequate FOBT | 3 months
  The investigators will register the number of cases in each arm where the result of the FOBT is unknown because the test was inadequate, that is, the test could not be read.
Proportion of positive FOBT referred for colonoscopy | 3 months
  The investigators will calculate the proportion of participants with a positive result in the FOBT that were referred to receive colonoscopy.
Implementation outcomes according to the RE-AIM framework | 3 months
  Implementation outcomes are: Reach, Effective implementation, adoption, implementation fidelity and maintenance

CONTACTS AND LOCATIONS:
Overall Officials: Vilma Irazola, Principal Investigator — Institute for Clinical Effectiveness and Health Policy
Locations (1):
- Ministry of Health, Mendoza, Argentina

REFERENCES:
- [Derived] Irazola V, Santero M, Sanchez M, Tristao I, Ruiz JI, Spira C, Ismael J, Cavallo AS, Gutierrez L, Mazzaresi Y, Nadal AM, Garcia Elorrio E; CCR Trial development group. Quality improvement intervention to increase colorectal cancer screening at the primary care setting: a cluster-randomised controlled trial. BMJ Open Qual. 2023 Jun;12(2):e002158. doi: 10.1136/bmjoq-2022-002158. PMID 37339820